CLINICAL TRIAL: NCT02885064
Title: Shifts in the Oral Biofilm of Patients With Known Oral Health Risk Factors
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1624
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2021-12-14 (Actual); Status verified 2021-04

CONDITIONS: Dental Caries; Gingivitis
MeSH Terms: conditions — Dental Caries; Gingivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bacteria isolated from plaque and saliva; human genome
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is observational only and is intended to evaluate changes in the makeup and function of bacteria naturally present in the mouth during treatment with braces to straighten teeth.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II (ASA I is a healthy patient, ASA II is patient with minor systemic disease)
* Patient must be receiving orthodontic treatment at the University of North Carolina School of Dentistry and not yet be in active treatment

Exclusion Criteria:

* Patients who have used antibacterial therapy in the past 3 months
* Patients who report current smoking
* ASA III or above (Patients with severe systemic diseases)

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients entering and then undergoing orthodontic treatment
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Change in Shannon diversity index from Baseline to Month 6 | Baseline, Month 6
Change from Baseline to Month 6 in Clusters Of Orthologous Groups of proteins | Baseline, Month 6

SECONDARY OUTCOMES:
Change in gingival index | Baseline, Month 6
Change in decalcification index | Baseline, Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Laura Jacox, DMD, PhD, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided